CLINICAL TRIAL: NCT01365871
Title: Pain Relief With Local Anesthetic at Time of Prostate Biopsy: Comparing Apical and Basal Injection Versus Basal Injection Alone
Brief Title: CREMS Prostate Biopsy Pain Relief Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Dr. Ants Toi, University Health Network, Toronto, Ontario, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TOI-CREMS
Record Dates: First submitted 2011-05-27; First posted 2011-06-03 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Pain
Keywords: prostate biopsy; pain
MeSH Terms: conditions — Pain | interventions — Anesthetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- basal injection (Active Comparator): basal injection of anesthetics
  Interventions: Procedure: anesthetics injection
- basal + apical injection (Active Comparator): basal + apical injection of anesthetics
  Interventions: Procedure: anesthetics injection

INTERVENTIONS:
Procedure: anesthetics injection — Basal injection of anesthetics or basal + apical injection of anesthetics.

SUMMARY:
The current standard for pain relief during prostate biopsy is the injection of local anesthetic agents into or around the prostate at various sites including apex, base, lateral aspects and into the prostate itself. Despite such anesthetic injection, some men still experience severe pain and often at the base of the penis. The study audits current practices comparing the degree of pain relief provided by injection at basal versus basal+apical sites. All these injection sites are standard practice at our hospital.

ELIGIBILITY:
Inclusion Criteria:

* Men who come for prostate biopsy

Exclusion Criteria:

* Men who are unwilling or unable to consent and fill in the forms

Min Age: 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pain scores comparing two groups. | post prostate biopsy procedure up to 6 months
  Pain questionnaires will be asked to filled in before the procedure, within 20 minutes of the procedure, at 2-4 weeks and at 6-month post procedure.

SECONDARY OUTCOMES:
Incidence of side effects and complications. | post prostate biopsy procedure up to 6 months
  Questionnaires will be asked to filled in to assess side effects and complications at 2-4 weeks and at 6-month post procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Ants Toi, MD, Principal Investigator — University Health Network, Toronto